CLINICAL TRIAL: NCT02862470
Title: Anaplastic Thyroid Cancer and Follicular Thyroid Cancer-derived Exosomal Analysis Via Treatment of Lovastatin and Vildagliptin and Pilot Prognostic Study Via Urine Exosomal Biological Markers in Thyroid Cancer Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201512110RINB
Record Dates: First submitted 2016-07-27; First posted 2016-08-11 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Thyroid Cancer
Keywords: Lovastatin; Vildagliptin; Exosome; Anaplastic thyroid cancer; Proteomics; Urine; Biological marker
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Carcinoma, Anaplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators expected to enroll 30 patients with papillary, follicular or anaplastic thyroid cancer, and collect their urine samples before operation, immediately after operation, post-operative 3, 6 12 months. The investigators will analyze the urine exosomal proteins and probable biological markers. The investigators hope to find the prognostic biological markers via this prospective study. The investigators further hope to find newly therapeutic mechanism and medications for such patients with poorly-differentiated or anaplastic thyroid cancer.

DETAILED DESCRIPTION:
Although papillary and follicular thyroid cancers are low-grade endocrine malignancy, they were fatal if the cancer cells were poorly-differentiated or anaplastic change. Prior researches indicated that one-third well-differentiated thyroid cancers could transform to poorly-differentiated patterns, even to be anaplastic thyroid cancer (ATC), a fatal malignancy, and no effective therapeutic strategies was noted, including surgical intervention, chemotherapy and radiotherapy. The poorly-differentiated or anaplastic change of thyroid cancer cells proliferates rapidly and always invades local tissues with distant metastasis. Cellular de-differentiation is the most pivotal cause for malignant transformation and invasion. De-differentiation usually in papillary thyroid cancer and follicular thyroid cancer, and definitely in ATC. The Poorly-differentiated thyroid cancer cell will rapidly proliferate and metastasize. The poorly-differentiated tumor cells lost apoptotic mechanism with de-differentiation, and such phenomenon is fatal for such patients. The investigators started research of thyroid cancer since 1999, and the investigators initially found TNF-α could induce cyto-morphological re-differentiation of thyroid cancer cells. Later, the investigators further found Lovastatin could induce re-differentiation of anaplastic thyroid cancer (ATC) cells in 25μM, but induce apoptosis in 50μM, in 2001. In 2006, the investigators designed nude mice model, and found tumor will shrink via treatment of Lovastatin in 5 or 10 mg/kg/day, but tumor will proliferate significantly in 1 mg/kg/day. The investigators called this phenomenon as "Duality effects" of statins. In 2012, the investigators found FLOT1 and transketolase (TKT) as important regulatory factor of re-differentiation and proliferation in ATC cells, respectively. The investigators also found that inhibition of Dipeptidyl peptidase-4 (CD26) will influence proliferation of ATC cells. Exosomes are nanovesicels secreted into extracellular environments. A growing evidence suggests theat exosomes could be used as biomarkers to be the diagnosis and prognosis of malignant tumors. Exosomes are 50-100 nm diameters, and correspond to the intrluminal vesicles of endosomal multivesicular bodies. Because of their cellular orgins, exosomes have specific protein markers, like CD63, CD9, CD81 and heat shock protein (HSP). Urine was used to be the biosamples in the past five years in baldder cancer, prostate cancer, breast cancer and ovarian cancer. Urine sample is usually easy to obtain and non-invasive. Exosomes secreted by cells could micro-molecularly transfer messages between cells and to be biological markers of cancer. The investigators now found Vildagliptin and Lovastatin could influence tumor cells survival via exosomal proteins. For patients of thyroid cancer, the investigators could obtain the urine samples without invasive procedures. Furthermore, the investigators could find the biological markers and therapeutic targets via the exosomal expression in urine. On the continuing basis of ATC cells culture experiments, the investigators expected to enroll 30 patients with papillary, follicular or anaplastic thyroid cancer, and collect their urine samples before operation, immediately after operation, post-operative 3, 6 12 months. The investigators will analyze the urine exosomal proteins and probable biological markers. The investigators hope to find the prognostic biological markers via this prospective study. The investigators further hope to find newly therapeutic mechanism and medications for such patients with poorly-differentiated or anaplastic thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with thyroid papillary, follicular and anaplastic thyroid cancer

Exclusion Criteria:

* Thyroid papillary, follicular and anaplastic thyroid cancer with prior operation, chemotherapy, or isotope treatment, or target therapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll the newly diagnosed patients with thyroid papillary, follicular and anaplastic thyroid cancer. After signing inform consent, the investigators will collect their urine samples before operation, immediately after operation, post-operative 3, 6 12 months (5 times in one patient).
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Prognostic biological markers via this prospective study. | 2 years
  Our study was designed as prospective pattern, and the investigators enrolled new thyroid cancer with follow-up, then detect urine exosome and proteins. The investigators try to find the correlation of outcome ( including recurrence, lymph nodes metastasis..) together with unknown/fresh biomarkers in this study and time-dependent manner.

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-YUAN WANG, Doctor, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang TY, Wang CY, Chen KY, Huang LT. Urinary Exosomal Thyroglobulin in Thyroid Cancer Patients With Post-ablative Therapy: A New Biomarker in Thyroid Cancer. Front Endocrinol (Lausanne). 2020 Jun 16;11:382. doi: 10.3389/fendo.2020.00382. eCollection 2020. PMID 32612576